CLINICAL TRIAL: NCT06486324
Title: Investigation of the Effects of Rapid Maxillary Expansion With Locked Modified Acrylic Bonded Appliance on Dentofacial Structures in Mixed Dentition
Brief Title: Effects of Asymmetric Rapid Maxillary Expansion on Dentoskeletal Structures in Mixed Dentition
Acronym: ARME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Irgin (Other)
Collaborators: Selcuk University (Other)
Responsible Party: Sponsor-Investigator, Celal Irgin, Assistant Professor, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 08102026
Record Dates: First submitted 2024-06-18; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Maxillary Anomaly; Asymmetric Maxillary Arch (Disorder); Cross Bite
Keywords: True unilateral posterior crossbite; Asymmetric maxillary expansion; Mixed dentition
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: Split-mouth model. The crossbite side of the patients was assigned as the treatment group, while the normal bite or non-crossbite side of the same patients was assigned as the positive control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Crossbite Side
  Interventions: Device: A locked modified acrylic bonded rapid maxillary expansion appliance (ARME)
- Positive Control Group (Experimental): Non-cossbite Side
  Interventions: Device: A locked modified acrylic bonded rapid maxillary expansion appliance (ARME)

INTERVENTIONS:
Device: A locked modified acrylic bonded rapid maxillary expansion appliance (ARME) — asymmetric maxillary expansion
  Other Names: Narrow maxillary half intended for expansion or crossbite side
  Arms: Treatment Group
Device: A locked modified acrylic bonded rapid maxillary expansion appliance (ARME) — asymmetric maxillary expansion
  Other Names: Normal maxillary half or non-crossbite side
  Arms: Positive Control Group

SUMMARY:
The aim of this clinical trial was to determine the efficacy of a locked modified bonded acrylic rapid maxillary expansion appliance, also known as an asymmetric rapid maxillary expansion appliance (ARME), in patients with a true unilateral posterior crossbite resulting from transversal maxillary deficiency in the mixed dentition.

DETAILED DESCRIPTION:
A posterior crossbite (PCB) is defined as an abnormal transverse or inverse relationship between the posterior teeth and dentition of the upper and lower jaws. A full buccal segment PCB involves multiple teeth in the posterior dentition and usually represents a transverse size discrepancy between the maxillary and mandibular relationships. This discrepancy is often caused by narrow or underdeveloped transverse dimensions of the maxillary halves. The underlying etiology of PCBs includes congenital, developmental, traumatic, or iatrogenic causes. Since spontaneous correction of this malocclusion is not possible even if the etiological factors are eliminated, it should be treated with maxillary expansion as early as possible.

The PCBs may be seen a unilateral posterior crossbite (UPCB) or bilateral posterior crossbite during all periods of dentition. A UPCB can be described as a functional UPCB or true UPCB. A functional UPCB is usually associated with a lateral shift of the mandible toward the crossbite side during the transition of the mandible. On the other hand, true UPCB is less common than functional UPCB and is caused by the narrowing of one of the maxillary halves. Increasing the maxillary arch transverse dimension is the main goal in the treatment of PCB. Although bilateral maxillary expansion is usually used to symmetrically widen the maxillary arch and eliminate mandibular shift as a standard treatment model in functional PCB, asymmetrical or unilateral maxillary expansion is recommended to expand narrowed sections of the maxillary halves and prevent overexpansion of the non-crossbite side in the treatment of true UPCB. Therefore, several removable or fixed maxillary expansion appliances that are slowly or rapidly activated were modified to produce differential effects on posterior teeth.

This clinical trial was designed to expand the upper jaw asymmetrically, i.e. to prevent the normal side of the bite from expanding while expanding the narrow part of the upper jaw. For this purpose, a locking mechanism was added to a bonded rapid maxillary expansion (RME) appliance to support the lower posterior teeth on the normal side of the bite.The hypothesis tested in the study was whether the true unilateral posterior cross-bite in the mixed dentition period could be corrected with a locked modified bonded rapid maxillary expansion appliance used for asymmetric expansion.

Children aged between 7 and 10 years old with true unilateral posterior crossbite were enrolled in the study. The efficacy of the appliance was compared between the crossbite and non-crossbite sides in the patients included in the study. The crossbite side of the patients was assigned as the treatment group, while the normal bite or noncrossbite side was assigned as the positive control group. Thus, two groups were formed for the study, and the trial was conducted on these groups.In other words, the study was planned as a self-controlled study. A negative control group could not be formed due to ethical reason. The reason for this is that the transversal problem may negatively affect both the anterioposterior and vertical development of the jaws in patients of this age during the developmental period, and therefore it was deemed necessary to correct the cross-bite problem as soon as possible after it was detected.Therefore, the purpose of this study was to evaluate specific dentoskeletal changes induced by treatment with true UPCB in mixed dentition with asymmetric RME.

ELIGIBILITY:
Inclusion Criteria:

* mixed dentition
* true unilateral posterior crossbite
* erupted first permanent molars and incisors
* all deciduous canines and molars or no more than one missing deciduous molar
* no history of orthodontic treatment
* no systemic disease
* no pathological periodontal status
* no excessive gagging reflex.

Exclusion Criteria:

* poor oral hygiene
* caries

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Widths of skeletal structures | Before expansion (T1),through expansion completion,an average 1 month (T2),and through retention completion, an average 3 months (T3)
  The widths of the nasal cavity, maxilla and mandible were measured in millimetres on the frontal radiographs and these widths were also determined separately on both the crossbite and non-crossbite sides.This involved marking anatomical points (lateral piriform rim,jugale, gonial notch and Lo points on both sides of the face and crista galli, a single point) and drawing two reference lines.The horizontal reference line was drawn by connecting the Lo points on both sides.The perpendicular line drawn from the crista galli to the horizontal reference line was the midsagittal line, which divided the face into two separate halves.The distances between the inter lateral piriform points, the inter jugular points and the inter gonial points corresponded to the width of the nasal cavity, the maxillary width and the mandibular width, respectively.The distances between the anatomical points on one half of the face to the midsagittal line indicated the skeletal width on that side.
Skeletal maxillomandibular width ratios | Before expansion(T1),through expansion completion an average 1 month(T2),and through retention completion an average 3 months(T3)
  The skeletal maxillomandibular ratio was calculated by dividing the skeletal maxillary width by the skeletal mandibular width and multiplying the result by 100. This percentage was calculated separately for the crossbite and non-crossbite sides and also for the total maxillary and mandibular width.
Inclinations of upper and lower first molars | Before expansion(T1),through expansion completion an average 1 month(T2),and through retention completion an average 3 months(T3)
  The angle formed by the intersection of the horizontal reference line with the line indicating the axis of a molar tooth defines the angular inclination of the molar tooth. The line indicating the axis of a molar was defined by the line connecting the crest of the buccal tubercle of the tooth and the most external part of the buccal curvature of the crown on the frontal radiograph. The angular inclinations of the upper and lower first molars were measured in degrees on frontal radiographs.
Amount of movement of deciduous canines and first molars in the transversal plane on the crossbite and non-crossbite sides. | Before expansion(T1),through expansion completion an average 1 month(T2),and through retention completion an average 3 months(T3)
  The perpendicular distances of deciduous canines and permanent first molars on the crossbite and non-crossbite sides to the median plane (MP), which was established as the reference plane on the dental cast. Distance measurements of the teeth were made in millimeter and these measurements represent the amount of movement of the canines and molars in the transverse plane.
Intercanine and intermolar distance on dental cast | Before expansion(T1),through expansion completion an average 1 month(T2),and through retention completion an average 3 months(T3)
  The distance measurement between the deciduous canines in the transversal plane on the upper and lower dental casts (intercanine distance). The distance measurement between the permanent first molars in the transversal plane on the upper and lower dental casts (intermolar distance). Distance measurements of the teeth were made in millimeter.

SECONDARY OUTCOMES:
Position of the maxilla in the sagittal and vertical plane on lateral cephalometric radiography | Before expansion(T1),through expansion completion an average 1 month(T2),and through retention completion an average 3 months(T3)
  1) SNA angle:The angle formed between the anterior cranial base (SN plane) passing through the Sella (S) and Nasion (N) points and the NA plane passing through the N and A points.It shows the sagittal position of the maxilla in degrees.2)SV⊥A (mm): The perpendicular distance of point A to the Sella Vertical (SV) line. SV was constructed through the Sella, perpendicular to the SN plane. It gives the position of the maxilla in the sagittal direction in millimetres.3)SN-PP angle: The angle formed between the SN plane and the palatal plane (PP) passing through the anterior nasal spine (ANS) and posterior nasal spine (PNS).It shows the vertical position of the maxilla and maxillary rotation in degrees.4)SN⊥ANS (mm): The perpendicular distance of ANS to SN plane. It gives the position of the ANS in the vertical position in millimetres.5)SN⊥PNS (mm): The perpendicular distance of PNS to SN plane. It gives the position of the PNS in the vertical direction in millimetres.
Position of the mandibula in the sagittal and vertical plane on lateral cephalometric radiograph | Before expansion(T1),through expansion completion an average 1 month(T2),and through retention completion an average 3 months(T3)
  1. SNB angle:The angle formed between the anterior cranial base (SN plane) passing through the Sella (S) and Nasion (N) points and the NB plane passing through the Nasion and B points on lateral cephalometric radiography. It shows the sagittal position of the mandible relative to the anterior cranial base in degrees.
  2. SV⊥B (mm): The perpendicular distance of point B to the Sella Vertical line (SV). SV was constructed through the Sella, perpendicular to the SN plane. It gives the position of the mandible in the sagittal direction in millimetres.
  3. SN-MP angle: The angle formed between the anterior cranial base (SN plane) passing through the Sella (S) and Nasion (N) points and the mandibular plane (MP) (Gonion-Menton) on lateral cephalometric radiography. It gives information about mandibular vertical position and mandibular rotation in degrees.
Maxillomandibular relationship in the sagittal plane on lateral cephalometric radiograph | Before expansion(T1),through expansion completion an average 1 month(T2),and through retention completion an average 3 months(T3)
  ANB angle: The angle formed between the NA and NB planes. It shows the positions of the maxilla and mandible relative to each other in the sagittal direction in degrees.
Skeletal midface and lower face heights in vertical plane on lateral cephalometric radiograph | Before expansion(T1),through expansion completion an average 1 month(T2),and through retention completion an average 3 months(T3)
  1. N-ANS (mm): The distance between Nasion (N) and anterior nasal spine (ANS). It shows the skeletal midface height in millimetres.
  2. ANS-Me (mm): The distance between anterior nasal spine (ANS) and menton (Me). It shows the skeletal lower face height in millimetres.
Angulation and position of the upper central incisor on lateral cephalometric radiograph | Before expansion(T1),through expansion completion an average 1 month(T2),and through retention completion an average 3 months(T3)
  1. U1_SN°: The angle between the long axis of the upper central incisor (U1) and the anterior cranial base (SN plane). It shows the angulation of the upper central incisor relative to the anterior cranial base in degrees.
  2. SV⊥U1 (mm): The perpendicular distance of incisal edge of the upper central incisor (U1) to Sella Vertical (SV) line. It gives the position of the upper central incisor in the sagittal direction in millimetres.
Angulation and position of the lower central incisor on lateral cephalometric radiograph | Before expansion(T1),through expansion completion an average 1 month(T2),and through retention completion an average 3 months(T3)
  1. L1_MP°: The angle formed between the axis of the most anteriorly located central incisor tooth in the mandible (L1) and the mandibular plane (MP). It gives the angulation of lower central incisor in degrees.
  2. SV⊥L1 (mm): The perpendicular distance of incisal edge of lower central incisor to Sella Vertical (SV) line. It gives the position of the lower central incisor in the sagittal direction in millimetres.

CONTACTS AND LOCATIONS:
Overall Officials: Celal Irgın, Asst.Prof., Principal Investigator — Selcuk University

IPD SHARING:
Plan to Share IPD: No
The study will be made available for sharing as soon as it has been turned into an article.

REFERENCES:
- [Result] Toroglu MS, Uzel E, Kayalioglu M, Uzel I. Asymmetric maxillary expansion (AMEX) appliance for treatment of true unilateral posterior crossbite. Am J Orthod Dentofacial Orthop. 2002 Aug;122(2):164-73. doi: 10.1067/mod.2002.125563. PMID 12165770
- [Result] da Silva Filho OG, Boas MC, Capelozza Filho L. Rapid maxillary expansion in the primary and mixed dentitions: a cephalometric evaluation. Am J Orthod Dentofacial Orthop. 1991 Aug;100(2):171-9. doi: 10.1016/s0889-5406(05)81524-0. PMID 1867168
- [Result] Sari Z, Uysal T, Usumez S, Basciftci FA. Rapid maxillary expansion. Is it better in the mixed or in the permanent dentition? Angle Orthod. 2003 Dec;73(6):654-61. doi: 10.1043/0003-3219(2003)0732.0.CO;2. PMID 14719729